CLINICAL TRIAL: NCT04184674
Title: Impact of the Transpulmonary Pressure on Right Ventricle Function in Acute Respiratory Distress Syndrome
Acronym: VD-SDRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP191033; 2019-A02814-53 (Other: IDRCB number)
Record Dates: First submitted 2019-11-28; First posted 2019-12-03 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Acute Respiratory Distress Syndrome; Mechanical ventilation; Transpulmonary pressure; Right ventricle failure
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Acute Respiratory Distress Syndrome (Other): Children of more than one month of age and adults hospitalized in Intensive Care Unit for Acute Respiratory Distress Syndrome.
  Interventions: Other: Pneumotachograph; Other: Esophageal catheter; Other: Transthoracic and / or transesophageal cardiac ultrasound; Other: Electrical impedance tomography (EIT) for pediatric patients

INTERVENTIONS:
Other: Pneumotachograph — Measurements will be performed during the first three days of Acute Respiratory Distress Syndrome management :
  * The first measurement will be performed 5 minutes after the initial ventilator settings.
  * Measurements will be repeated systematically at 24 hours, 48 hours and 72 hours of evolution.
  * An additional measure will be performed at each positive end-expiratory pressure modification (maximum 5 measures).
Other: Esophageal catheter — Measurements will be performed during the first three days of Acute Respiratory Distress Syndrome management
  * The first measurement will be performed 5 minutes after the initial ventilator settings.
  * Measurements will be repeated systematically at 24 hours, 48 hours and 72 hours of evolution.
  * An additional measure will be performed at each positive end-expiratory pressure modification (maximum 5 measures).
Other: Transthoracic and / or transesophageal cardiac ultrasound — The right ventricle systolic function will be assessed thanks to a transthoracic cardiac ultrasound in children, and a transthoracic of a transesophageal cardiac ultrasound in adults :
  Measurements will be performed during the first three days of Acute Respiratory Distress Syndrome management :
  * The first measurement will be performed 5 minutes after the initial ventilator settings.
  * Measurements will be repeated systematically at 24 hours, 48 hours and 72 hours of evolution.
  * An additional measure will be performed at each positive end-expiratory pressure modification (maximum 5 measures).
Other: Electrical impedance tomography (EIT) for pediatric patients — For pediatric patients: measurements will be performed during the first three days of Acute Respiratory Distress Syndrome management.

SUMMARY:
Pulmonary distension induced by mechanical ventilation physiologically alters right ventricle pre and after-load, hence might lead to right ventricle failure. The hypothesis is that in Acute Respiratory Distress Syndrome, the occurence of a right ventricle failure under lung protective ventilation might :

i) be correlated to the transpulmonary pressure level, ii) lead to global heart failure, iii) and extremely result in poor outcome and death.

The primary objective is to test the impact of transpulmonary pressure on right ventricular function in Acute Respiratory Distress Syndrome in adults and children.

Secondary objectives are :

i) to compare thresholds of transpulmonary pressure associated with right ventricle failure between children and adults.

ii) to assess if there is an association between transpulmonary pressure and morbidity and mortality.

- For pediatric patients, a specific monitoring with electrical impedance tomography (EIT) will allow:

* To assess if the transpulmonary pressure is associated with the level of regional pulmonary overdistention (or collapse) on electrical impedance tomography.(EIT)
* To assess if there is an association between the occurrence of right ventricular failure, and distribution of ventilation on EIT.

DETAILED DESCRIPTION:
Acute Respiratory Distress Syndrome (ARDS) is an acute inflammatory lung injury associated with a high pulmonary vascular permeability, leading to acute respiratory failure. Positive pressure mechanical ventilation,improves survival but might lead to ventilator-induced lung injury (VILI) and right ventricular failure. This hemodynamic effect is more important when compliance is decreased, especially in ARDS.

The use of long protective ventilation (with low tidal volumes and low plateau pressures) has improved prognosis of ARDS in adult patients. However, tidal volume and plateau pressures do not always reflect the lung deformation and the stress induced by the ventilation; these variables depend on the characteristics of the patient's respiratory system. Therefore, management focuses on ventilation strategies according to these characteristics.

Among tools used to evaluate respiratory physiological parameters, the esophageal pressure measurement is easily feasible at the bedside, and well estimates pleural pressure and pulmonary distension. During invasive ventilation, transpulmonary pressure (PL) can be obtained with the difference between the airway pressure and the esophageal pressure. Calculation of transpulmonary pressure in ARDS allows optimal ventilator management of adult and children treated for ARDS.

Although individualized ventilation techniques have shown some benefits in ARDS, studies have failed to show that survival could be improved by such strategies. This lack of efficacy could be partly explained by the hemodynamic impact of ventilation-induced pulmonary distension. It therefore seems essential to combine a robust assessment of right ventricular function with measurements of transpulmonary pressure in order to know the real hemodynamic impact of positive pressure ventilation in ARDS in adults and children.

The primary objective is to test the impact of transpulmonary pressure on right ventricular functionin ARDS adults and children.

Secondary objectives are :

i) to compare thresholds of transpulmonary pressure associated to right ventricle failure between children and adults ii) to assess if there is an association between transpulmonary pressure and morbidity and mortality.

- For pediatric patients, a specific monitoring with electrical impedance tomography (EIT) will allow:

* To assess if the transpulmonary pressure is associated with the level of regional pulmonary overdistention (or collapse) on electrical impedance tomography.(EIT)
* To assess if there is an association between the occurrence of right ventricular failure, and distribution of ventilation on EIT.

ELIGIBILITY:
Inclusion Criteria:

* Patients over one month
* Patients with mild to severe ARDS (onset within 48 hours). ARDS definition will follow Berlin guidelines for adults, and Pediatric Acute Lung Injury Consensus Conference (PALICC) guidelines for children
* Signed consent

Exclusion Criteria :

* Neonates less than 28 days-old
* Pregnancy or breastfeeding
* Any contra-indication to esophageal manometry (less than one month esophagus surgery, bronchopleural or esotracheal fistula, latex allergy)
* No social care

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2022-06-11 (Actual); Study Completion 2022-06-11 (Actual)

PRIMARY OUTCOMES:
Right ventricle failure | Three days
  Right ventricle failure is defined, by ultrasound, as a composite criteria associating :
  * end-diastolic right ventricle/left ventricle area ratio > 0.6 and/or Acute Cor Pulmonale (assocation with a septal dyskinesia),
  * and/or a tricuspid annular plane systolic excursion < 1,6 cm (adults), z-score < -2 (children),
  * and/or a doppler-derived tricuspid lateral annular systolic velocity (S wave) < 10 cm/s,
  * and/or a two-dimensional Fractional Area Change (defined as end-diastolic area - end-systolic area)/end-diastolic area x100) < 35%,
  * and/or a peak right ventricle free wall 2D strain < -30% (adults), z-score < 2 (children).

SECONDARY OUTCOMES:
Airways pressure | Three days
  Airways pressure (Paw) will be measured in cmH2O thanks to a pneumotachograph connected to the ventilator.
Oesophageal pressure | Three days
  Esophageal pressure (Pes) will be measured in cmH2O thanks to an oesophageal balloon catheter introduced in the mid-esophagus of the patient and connected to a manometer.
Transpulmonary pressure calculation | Three days
  Measurements will be performed at different moments during the respiratory cycle: after an inspiratory pause to evaluate the tele-inspiratory transpulmonary pressure (PL-insp), and after an expiratory pause to evaluate the tele-expiratory transpulmonary pressure (PL-PEP ). The PL-insp will be calculated using the ratio between the elastance of the chest wall (Ecw) and of the respiratory system (Ers) thanks to this formula PL = Paw - Paw x (Ecw/Ers). The PL-exp will be calculated using the ratio between Paw et Pes (PL = Paw - Pes). Transpulmonary pressure will be expressed in cmH2O.
Vaso-Active Inotrope Score (VIS) | Three days
  Correlation between transpulmonary pressure and morbidity. Vaso-Active Inotrope Score is a hemodynamic score taking into account the cumulative doses of inotropic or vassopressive drugs. It is obtained thanks this calculation : VIS = dopamine dose (µg/kg/min) + dobutamine dose (µg/kg/min) + 100 x epinephrine dose (µg/kg/min) + 10 x milrinone dose (µg/kg/min) + 10000 x vasopressin dose (µg/kg/min) + 100 x norepinephrine dose (µg/kg/min). Its value ranges from zero, which is associated to a better outcome, to the maximum cumulative dose without any limit.
Duration of treatment with vasoactive or inotropic drugs | 3 months after hospitalization in Intensive Care Unit
  Number of days under vaso-active or inotropic drugs
Pediatric logistic organ dysfunction score | Three days
  Pediatric logistic organ dysfunction score is a specific pediatric multiple organ dysfunction score that includes 10 variables corresponding to 5 organ dysfunctions. Values extend from 0 (best outcome) to 33 (worst outcome).
Sepsis-related Organ Function Assessement score | Three days
  Sepsis-related Organ Function Assessement score is a multiple organ dysfunction score that includes several variables corresponding to 6 organ dysfunctions. Values extend from 0 (best outcome) to 24 (worst outcome).
Invasive and non invasive ventilation free days | 3 months after hospitalization in Intensive Care Unit
  Number of invasive and non invasive ventilation free days
Lung and Chest Wall compliance | Three days
  Lung and chest wall compliances (in mL/cmH2O) will be calculated thanks to the respective ratios tidal volume/(PL-insp - PL-PEP) and tidal volume/(Pes insp - Pes-PEP).
Length of hospitalization | 3 months after hospitalization in Intensive Care Unit
  Length of hospitalization in Intensive Care Unit and in hospital in days.
Mortality at 28 days | 28 days
  Death in Intensive Care Unit and at 28 days of hospitalization.
Mortality in Intensive Care Unit | 3 months after hospitalization in Intensive Care Unit
  Death in Intensive Care Unit.
Eletrical impedance tomography | 3 days
  Electrical impedance tomography will be monitored only in children. Several methods will be used and compared, based on e.g. pixel information of lung aeration, to assess end-expiratory lung volume (ELLV, in mL) and the distribution of ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Meryl Vedrenne-Cloquet, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Brigitte Fauroux, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - Hôpital Necker-Enfants Malades, Paris

REFERENCES:
- [Background] Vedrenne-Cloquet M, Petit M, Khirani S, Charron C, Khraiche D, Panaioli E, Habib M, Renolleau S, Fauroux B, Vieillard-Baron A. Impact of the transpulmonary pressure on right ventricle impairment incidence during acute respiratory distress syndrome: a pilot study in adults and children. Intensive Care Med Exp. 2024 Sep 27;12(1):84. doi: 10.1186/s40635-024-00671-2. PMID 39331249